CLINICAL TRIAL: NCT01801046
Title: HLA-mismatched Allogeneic Cellular Therapy (HMMACT) After Chemotherapy in High Risk Acute Myeloid Leukemia
Brief Title: Donor Stem Cell Transplant in Treating Patients With High Risk Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-11-8; NCI-2013-00447 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myeloid Leukemia in Remission; Childhood Acute Myelomonocytic Leukemia (M4); Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Mitoxantrone; Cytarabine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, G-PBSC) (Experimental): INDUCTION CHEMOTHERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-3 and cytarabine IV on days 1-7. HMMACT: Patients receive G-PBSC on day 9.
  Interventions: Drug: mitoxantrone hydrochloride; Drug: cytarabine; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Procedure: peripheral blood stem cell transplantation — Undergo HMMACT with G-PBSC
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects of donor stem cell transplant in treating patients with high risk acute myeloid leukemia. Giving low doses of chemotherapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells when they do not exactly match the patient's blood. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of cytarabine based chemotherapy and human leukocyte antigen (HLA)-mismatched allogeneic cellular therapy (HMMACT) in patients with high risk acute myeloid leukemia (AML), with feasibility measured by induction mortality (IM) and complete response rate.

SECONDARY OBJECTIVES:

I. To obtain preliminary estimates of clinical outcome following cytarabine based chemotherapy and HMMACT in patients with high risk AML, as measured by event free survival (EFS) and overall survival (OS).

II. To further evaluate the safety outcomes of induction and consolidation of cytarabine and HMMACT in terms of serious infections (grade 4), time to recovery of absolute neutrophil counts and platelets and incidence of graft versus host disease (GvHD).

III. To further evaluate the feasibility of this approach in terms of identifying a suitable donor in this elderly population.

IV. To compare in preliminary manner the clinical outcomes of cytarabine and HMMACT in patients with high risk AML as measured by complete response rate (CRR), event free survival (EFS) and overall survival (OS) by donor/recipient HLA-C1 vs C2 pairs.

V. To characterize in a preliminary manner, the numbers of suppressor regulatory T cells (Tregs), T helper 17 cells (Th17), and cytotoxic T cells during pre and post HMMACT treatment, and with clinical outcomes in leukemia.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive mitoxantrone hydrochloride intravenously (IV) on days 1-3 and cytarabine IV on days 1-7.

HMMACT: Patients receive filgrastim (G-CSF) mobilized peripheral blood stem cells (G-PBSC) on day 9. After completion of study treatment, patients are followed up monthly for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically and cytological confirmed acute myeloid leukemia, high risk AML defined as:

  * Age > 60, or
  * Presence of complex cytogenetic abnormalities (with > 3 cytogenetic abnormalities), del (7q, -5, -7), t(9,22), 11q(23) or high risk mutations by FISH eg MLL, FLT-3 +
  * Secondary AML, or
  * A white blood cell count of > 50 x10^9/L
* Patients must be medically ineligible for allogeneic stem cell transplant (alloSCTx) or not have a known fully HLA matched sibling for planned sibling transplant.
* Patients must have measurable or evaluable disease
* Diagnosis of AML according to World Health Organization (WHO) diagnostic criteria (at least 20% blasts in the peripheral blood or bone marrow), with French-American-British Cooperative group (FAB) classification other than M3 (acute promyelocytic leukemia), documented by bone marrow aspiration and biopsy performed within 14 days prior to administration of 1st dose of remission induction chemotherapy; if a bone marrow aspirate and biopsy were obtained within 28 days prior to the first dose of remission induction therapy then these tests may be submitted for review at University of Southern California (USC) and a repeat screening bone marrow does not need to be conducted;

  * Cohort A: newly diagnosed AML, no prior cytotoxic chemotherapy
  * Cohort B: newly diagnosed AML, failed to achieve Complete remission (CR) with single standard Induction chemo.
* Patient has at least one medically fit family member expected to be HLA mismatched at 1-9/10; more commonly and preferred: 4-6/10 loci (parent, sibling, niece/nephew, etc but adult children preferred)
* Absolute neutrophil count (ANC) > 1500, unless due to direct bone marrow involvement of disease
* Platelets > 75,000, unless due to direct bone marrow involvement of disease
* Hemoglobin > 8.0 gm/dL, transfusion allowed
* Serum creatinine < 2.0 x the upper limits of institutional normal (ULN)
* Total bilirubin < 1.5 x the upper limits of institutional normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT )< 2.5 x the upper limits of institutional normal (=< 5 x ULN for patients with liver involvement of leukemia)
* Cardiac left ventricular ejection fraction (LVEF) > 45%
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Estimated survival of at least 3 months
* Patients must be able to understand and agree to sign an Institutional Review Board (IRB)-approved informed consent form
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study, and for two months after study participation
* DONOR: Donor screening; all donors will meet the standard blood donor criteria established by the participating local blood center, American Association of Blood Banks (AABB)
* DONOR: Donors will be selected from among the subject's relatives, adult children preferred
* DONOR: Infectious disease testing will be done per Hemacare policy and AAAB guidelines
* DONOR: Donor and intended recipient red cell type and compatibility will be determined
* DONOR: Donors will be pre-selected on the basis of HLA haploidentity
* DONOR: If patient is cytomegalovirus (CMV)-negative, donors who are CMV-negative will be preferred; CMV serology of the donor will be tested prior to the allogeneic cell donation; donations from CMV-positive donors to CMV-negative recipients will be given if no CMV negative donor is available, and CMV surveillance and pre-emptive treatment given

Exclusion Criteria:

* Cohort A: Patients who have received prior cytotoxic chemotherapy, such as anthracyclines and cytarabine not permitted; but prior treatment with demethylating agents (azacytidine or decitabine, lenalidomide, etc) ALLOWED.
* Cohort B: Patients who have received prior fludarabine, clorarabine or drugs known to target T cells not permitted; but prior standard induction with anthracylines and cytarabine ALLOWED including after demethylating agents.
* Have uncontrolled systemic infections, coagulation disorders, or other major medical illnesses of the cardiovascular or respiratory systems
* Pregnant and/or lactating
* Patients who have had non-biopsy surgery in the last 10 days
* Active central nervous system (CNS) disease; patients with previously treated leptomeningeal disease without evidence of remaining leukemia cells by spinal fluid will be eligible
* Known active autoimmune disorder
* Known to be human immunodeficiency virus (HIV)-positive or have active hepatitis B or C
* Patients concurrently taking the following drugs are excluded: mycophenolate, cyclosporine, prednisone > 20mg/day, or immunosuppressive agents
* DONOR: Personal or family history of severe sickle cell disease or variant (unless donor has tested negative); testing for the presence of hemoglobin S is not required
* DONOR: Positive infectious disease test as dictated by blood collection center's standard operating procedure (SOP)
* DONOR: Current uncontrolled hypertension
* DONOR: Diabetes mellitus
* DONOR: Active peptic ulcer disease
* DONOR: Pregnant or breast-feeding
* DONOR: Currently taking lithium therapy
* DONOR: History of autoimmune disease
* DONOR: History of coronary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Induction mortality | Up to 8 weeks
Complete remission rate (complete remission [CR] or incomplete remission [CRi]) | Up to 3 years
  Exact 95% confidence intervals will be constructed.

SECONDARY OUTCOMES:
Occurrence of serious infections (grade 4) assessed using National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) v4.0 | Up to 3 years
  Will be summarized in terms of type, severity, attribution, time of onset, duration, reversibility, and outcome.
Time to recovery of absolute neutrophil counts (ANC) | From stem cell infusion to the first of 3 consecutive days in which the ANC is more than 0.5 x 10^9/L, assessed up to 3 years
  Will be summarized using cumulative incidence curves.
Time to recovery of platelets | From stem cell infusion until the first of 3 consecutive days in which the platelet count is more than 30 x 10^9/L, assessed up to 3 years
  Will be summarized using cumulative incidence curves.
Incidence of GvHD | Up to 3 years
  Will be reported in terms of grade, site, and time of onset (for acute GvHD) and whether limited or extensive, and time of onset (for chronic GvHD).
Estimate of clinical outcome as measured by event free survival (EFS) | From the start of induction until documentation of failure to achieve a CR or CRi during induction, initiation of a salvage therapy, disease recurrence/progression (after induction), or death due to any cause, assessed up to 2 years
  Kaplan-Meier plots will be used to summarize the EFS observed in this series. The proportion of patients alive and in continuous complete remission will be estimated at 6, 12, 18, and 24 months. 95% intervals will be constructed.
Estimate of clinical outcome as measured by overall survival (OS) | From the start of induction until death due to any cause, assessed up to 2 years
  Kaplan-Meier plots will be used to summarize the OS observed in this series. The proportion of patients alive will be estimated at 6, 12, 18, and 24 months. 95% intervals will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mohrbacher, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States